CLINICAL TRIAL: NCT05506969
Title: Phase 2, Randomized, Active-Controlled, Observer-Blinded, Multicenter Trial of the Immunogenicity, Safety, and Tolerability of rF1V Vaccine With CpG 1018® Adjuvant Compared With rF1V Vaccine in Adults 18 to 55 Years of Age
Brief Title: Trial of the Immunogenicity, Safety, and Tolerability of rF1V Vaccine With CpG 1018® Adjuvant Compared With rF1V Vaccine in Adults 18 to 55 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: DV2-PLG-01
Record Dates: First submitted 2022-08-10; First posted 2022-08-18 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Plague, Pneumonic; Plague; Vaccine-Preventable Diseases
MeSH Terms: conditions — Plague; Vaccine-Preventable Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- rF1V-1018 co-administered (rF1V vaccine and CpG 1018® adjuvant co-administered) (Experimental): Co-administration of rF1V vaccine and CpG 1018® adjuvant administered as 2 injections
  Interventions: Biological: rF1V-1018
- rF1V-bedside mix (rF1V vaccine and CpG 1018® adjuvant bedside mix) (Experimental): Bedside mix of rF1V vaccine and CpG 1018® adjuvant administered administered as 2 injections
  Interventions: Biological: rF1V-1018
- rF1V vaccine only (Experimental): rF1V vaccine administered as 3 injections
  Interventions: Biological: rF1V vaccine

INTERVENTIONS:
Biological: rF1V-1018 — rF1V vaccine and CpG 1018® adjuvant
  Arms: rF1V-1018 co-administered (rF1V vaccine and CpG 1018® adjuvant co-administered); rF1V-bedside mix (rF1V vaccine and CpG 1018® adjuvant bedside mix)
Biological: rF1V vaccine — rF1V vaccine
  Arms: rF1V vaccine only

SUMMARY:
Phase 2, Randomized, Active-Controlled, Observer-Blinded, Multicenter Trial of the Immunogenicity, Safety, and Tolerability of rF1V Vaccine with CpG 1018® Adjuvant Compared with rF1V Vaccine in Adults 18 to 55 Years of Age

DETAILED DESCRIPTION:
Phase 2, randomized, active-controlled, observer-blind, multicenter trial of the immunogenicity, safety, and tolerability of rF1V vaccine with CpG 1018® adjuvant (rF1V-1018) compared with rF1V vaccine alone in adults. Approximately two hundred healthy adults 18 to 55 years of age will be enrolled to compare a two-dose regimen of rF1V-1018 with a three-dose regimen of rF1V vaccine alone. The study will be conducted in 2 parts (Part 1 and Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 55 years
* Healthy participants or participants with pre-existing medical conditions who are in a stable medical condition.

Pre-existing stable medical condition means a subject who: has full capacity of daily activity and no major medication modification within 3 months prior to Day 1; has not undergone surgical or minimally-invasive intervention or had any hospitalization/emergency room visit for the specific medical condition.

* Able to comply with the protocol schedule and procedures.
* Able and willing to provide written informed consent
* If female of child-bearing potential and heterosexually active, has practiced adequate contraception for 28 days prior to vaccination and has negative pregnancy tests just prior to vaccination and has agreed to continue adequate contraception until 28 days after last study injection. Adequate contraception is defined as a contraceptive method with a failure rate of < 1% per year when used consistently and correctly and, when applicable, in accordance with the product label. Examples include the following:

  * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, or transdermal
  * Progestin-only hormonal contraception associated with inhibition of ovulation: oral, injectable, or implantable
  * Intrauterine device (IUD) with or without hormonal release
  * Vasectomized partner, provided he is the subject's sole partner and that he has received a medical assessment of the surgical success
  * Credible self-reported history of heterosexual abstinence for at least 28 days prior to vaccine administration
  * Female partner

Exclusion Criteria:

* A history of plague disease or have previously received any plague vaccine.
* Active tuberculosis or other systemic infectious process.
* History of human immunodeficiency virus (HIV), hepatitis B (HBV) or hepatitis C (HCV) infection, or positive test for antibody to HIV, HBV, or HCV
* History of autoimmune disorder
* History of sensitivity to any component of study vaccines
* Body mass index ≥ 30 kg/m2
* Has received the following prior to the injection:
* 14 days:
* COVID-19 vaccine
* Any inactivated vaccine
* 28 days:
* Any live vaccine
* Systemic corticosteroids (more than 3 consecutive days) or other immunomodulators or immunomodulators immune suppressive medication, with the exception of inhaled steroids
* Any other investigational medicinal agent
* 90 days:
* Immunoglobulins or any blood products
* Granulocyte or granulocyte-macrophage colony-stimulating factor
* Antisense oligonucleotides
* Drugs/investigational agents with very long half-lives (defined as ≥ 60 days)
* At any time: DNA plasmids or other genetic therapy intended to integrate permanently into host cells
* If female is pregnant (known before or established at the time of screening), breastfeeding, or planning a pregnancy
* Is undergoing chemotherapy or expected to receive chemotherapy during the study period; has a diagnosis of cancer within the last 5 years other than squamous cell or basal cell carcinoma of the skin
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Oral temperature >100.0°F at the time of vaccine administration.
* History of acute myocardial infarction (AMI) or documented coronary artery disease (CAD)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2024-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Janssen, MD, Study Chair — Dynavax Technologies Corporation
Locations (6):
- United States (6):
  - Optimal Research Alabama, Huntsville, Alabama
  - Optimal Research California, San Diego, California
  - Optimal Research Florida, Melbourne, Florida
  - Optimal Research Illinois, Peoria, Illinois
  - Optimal Research Maryland, Rockville, Maryland
  - Optimal Research Texas, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- rF1V-1018 Co-Administered: rF1V vaccine and CpG 1018® adjuvant administered on Days 1 and 29, and 2 injections of placebo administered on Day 183
- rF1V-1018 Bedside Mix: Bedside mix of rF1V vaccine and CpG 1018® adjuvant administered on Days 1 and 29, and 2 injections of placebo administered on Day 183
- rF1V Vaccine Only: rF1V vaccine administered on Days 1, 29, and 183
Period: Overall Study
Arm/Group | rF1V-1018 Co-Administered | rF1V-1018 Bedside Mix | rF1V Vaccine Only
Started | 21 | 90 | 89
Completed | 18 | 81 | 77
Not Completed | 3 | 9 | 12

BASELINE CHARACTERISTICS:
Population: Safety analysis population: All participants who received at least 1 study injection and had any post-baseline safety data
Groups:
- Total: Total of all reporting groups
Arm/Group | rF1V-1018 Co-Administered | rF1V-1018 Bedside Mix | rF1V Vaccine Only | Total
Number analyzed (Participants) | 21 | 90 | 89 | 200
Age, Customized [Mean (Standard Deviation); unit: Years]
  Mean (SD) | 39.1 (8.17) | 40.0 (9.2) | 37.9 (9.91) | 39.0 (9.76)
Age, Customized [Count of Participants; unit: Participants]
  18-39 | 12 | 42 | 46 | 100
  40+ | 9 | 48 | 43 | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 34 | 36 | 79
  Male | 12 | 56 | 53 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 8 | 10 | 18
  Not Hispanic or Latino | 21 | 77 | 77 | 175
  Unknown or Not Reported | 0 | 5 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 62 | 62 | 138
  Black or African American | 4 | 19 | 20 | 43
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 1 | 2 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 2 | 3
  Other | 1 | 5 | 3 | 9
Body mass index [Mean (Standard Deviation); unit: (kg/m^2)] | 26.5 (2.46) | 25.9 (3.04) | 25.5 (3.16) | 25.8 (3.04)

OUTCOME MEASURES:

1. Primary Outcome: Rates of Reactogenicity and Safety
Description: Rates of solicited local and systemic post-injection reactions, and AEs, severe AEs, SAEs, AESIs, and deaths
Time Frame: Day 1 to Week 56
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | rF1V-1018 Co-Administered | rF1V-1018 Bedside Mix | rF1V Vaccine Only
Number analyzed (Participants) | 21 | 90 | 89
Participants
  Local Reactions | 16 | 67 | 57
  Severe Local Reactions | 0 | 0 | 2
  Systemic Reactions | 13 | 60 | 42
  Severe Systemic Reactions | 0 | 2 | 0
  At least 1 Unsolicited AE | 7 | 27 | 28
  Severe (Grade 3 or 4) AEs | 2 | 1 | 5
  SAEs | 1 | 0 | 3
  AESIs | 1 | 0 | 1
  Deaths | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Participants were followed for post-injection local and systemic reaction for 7 days post each injection and for AEs, SAEs, and imAESIs through Day 393 (Week 56).
Arm/Group | rF1V-1018 Co-Administered | rF1V-1018 Bedside Mix | rF1V Vaccine Only
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/90 | 1/89
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/90 | 3/89
Other Adverse Events (participants affected / at risk) | 18/21 | 77/90 | 69/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rF1V-1018 Co-Administered (N=21) | rF1V-1018 Bedside Mix (N=90) | rF1V Vaccine Only (N=89)
Cor Pulmonale Acute (Cardiac disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0 | 0
Complicated Appendicitis (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rF1V-1018 Co-Administered (N=21) | rF1V-1018 Bedside Mix (N=90) | rF1V Vaccine Only (N=89)
Chills (General disorders) | 3 | 13 | 14
Diarrhoea (Gastrointestinal disorders) | 7 | 15 | 12
Fatigue (General disorders) | 10 | 43 | 30
Headache (Nervous system disorders) | 8 | 34 | 25
Injection Site Pain (General disorders) | 16 | 66 | 56
Injection Site Pruritus (General disorders) | 2 | 17 | 13
Malaise (General disorders) | 6 | 25 | 21
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 23 | 22
Nausea (Gastrointestinal disorders) | 4 | 13 | 12
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT05506969/Prot_002.pdf
  • Statistical Analysis Plan (2024-06-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT05506969/SAP_003.pdf